CLINICAL TRIAL: NCT06395246
Title: The Usefulness of Circulating Microvesicles (host and Bacterial) in Regulating Metabolic Homeostasis in Obesity Randomized Study of Parallel Arms in Obese Patients Undergoing Caloric Restriction Diet Vs. Early Time-restricted Eating
Brief Title: Circulating Microvesicles Regulating Metabolic Homeostasis in Obesity After Caloric Restriction Programs
Acronym: TREV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Investigacio Sanitaria Pere Virgili (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI23/01133
Record Dates: First submitted 2024-04-24; First posted 2024-05-02 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Obesity
Keywords: obesity; extracellular vesicles; incretins; bile acids; short-chain fatty acids; time-restricted feeding; caloric restriction; brown fat
MeSH Terms: conditions — Obesity; Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: Randomized parallel-arm design (n=40) with consecutive 1:1 allocation to either a continuous calorie restriction diet (n=20) for a healthy Mediterranean diet or an early time-restricted eating protocol + continuous caloric restriction (n=20) over 12 weeks.
Who Masked: Investigator, Outcomes Assessor
Masking Description: triple-blind: participants, intervention researchers - except for the nutritionist in charge of diet and lifestyle counseling - and data analysts will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continuous caloric restriction (Active Comparator): Continuous calorie restriction diet based on healthy Mediterranean diet recommendations
  Interventions: Behavioral: Active Comparator: Continuous calorie restriction
- eTRE (Experimental): early (morning) time-restricted eating (eTRE) plus continuous caloric restriction diet based on healthy Mediterranean diet recommendations
  Interventions: Behavioral: eTRE

INTERVENTIONS:
Behavioral: Active Comparator: Continuous calorie restriction — Individualized continuous calorie restriction diet based on healthy Mediterranean diet recommendations aiming to achieve at least a 5% weight loss at the end of the intervention
  Arms: Continuous caloric restriction
Behavioral: eTRE — early (morning) time-restricted eating pluss individualized continuous calorie restriction diet based on healthy Mediterranean diet recommendations aiming to achieve at least a 5% weight loss at the end of the intervention
  Arms: eTRE

SUMMARY:
The main aim of the present study is to evaluate the effectiveness of two dietary protocols: Daily Caloric Restriction (DCR) and Early Time-Restricted Feeding + DCR (eTRE) on metabolic homeostasis and the influence of circulating extracellular vesicles (EVs) as inter-organ communication elements in obese patients.

DETAILED DESCRIPTION:
The specific objectives are:

1. To assess the effect of two dietary protocols on weight loss and metabolic benefits in non-morbidly obese subjects.
2. Influence of both protocols on energy signaling metabolites and the dynamics of enteroendocrine hormones.
3. Define the "digital footprint" of EVs as inter-organ communication elements influencing metabolic status in obese subjects.

The study design comprises a randomized parallel-arm design (n=40) with consecutive 1:1 allocation to a calorie restriction protocol for a healthy Mediterranean diet under Daily Caloric Restriction (DCR) (n=20) or an eTRE protocol (n=20) for 12 weeks. Clinical and analytical variables, adherence, satiety, chronotype, and brown fat content will be determined before and at the end of the follow-up. Derivatives of intestinal microbiota, short-chain fatty acids, bile acids, and circulating metabolites derived from host intermediary metabolism will be assessed through metabolomics. Glucagon-like peptide 1 (GLP1) and gastric inhibitory polypeptide (GIP) dynamics after a standard meal test. Metagenomics. Bioenergetic analysis of PBMC by SeaHorse. Total EV miRNA profile. Isolation of host and bacterial EVs. Characterization of the protein cargo of host and bacterial EVs.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 70 years old.
2. BMI ranges between 27 and 40 kg/ m2.
3. Absence of underlying pathology in medical and physical examination, except for those related to excess weight.
4. Signature of the informed consent for participation in the study.

Exclusion Criteria:

1. Serious systemic disease not related to obesity, such as cancer, kidney or severe liver disease.
2. Systemic diseases with intrinsic inflammatory activity (autoimmune diseases such as rheumatoid arthritis and asthma).
3. Pregnancy and lactation.
4. Vegetarians or subjects subjected to an irregular diet.
5. Patients with severe eating disorders.
6. Patients with clinical symptoms and signs of infection in the previous month.
7. Patients with chronic anti-inflammatory steroid treatments and/or nonsteroidal anti-inflammatory drugs.
8. Recent antibiotic treatment.
9. Uncontrolled alcoholism or drug abuse.
10. Rotating or nocturnal shift workers.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Anthropometric measurements (I) | Before and after (12 weeks) of the intervention
  Changes in weight (kg)
Anthropometric measurements (II) | Before and after (12 weeks) of the intervention
  Changes in body mass index (kg/m^2);
Anthropometric measurements (III) | Before and after (12 weeks) of the intervention
  Changes waist circumference (cm)
Anthropometric measurements (IV) | Before and after (12 weeks) of the intervention
  Changes hip circumference (cm)
Anthropometric measurements (V) | Before and after (12 weeks) of the intervention
  Changes neck circumference (cm)
Body composition (I) | Before and after (12 weeks) of the intervention
  Changes in fat body mass (kg); assesed by bioimpedance monitoring device (Seca®)
Body composition (II) | Before and after (12 weeks) of the intervention
  Changes in lean body mass (kg); assesed by bioimpedance monitoring device (Seca®)
Body composition (III) | Before and after (12 weeks) of the intervention
  Changes visceral adipose tissue (L); assesed by bioimpedance monitoring device (Seca®)
Brown fat | Before and after (12 weeks) of the intervention
  Changes in brown fat volume (cm3); assessed by magnetic resonance image (MRI)

SECONDARY OUTCOMES:
Gut and host microbiota-derived metabolites (I) | Before and after (12 weeks) of the intervention
  Changes in circulating short-chain fatty acids levels [µM]; assesed by Gas Chromatography-Tandem Mass Spectrometry (GC-MS/MS)
Gut and host microbiota-derived metabolites (II) | Before and after (12 weeks) of the intervention
  Changes in circulating bile acids levels [nM]; Liquid Chromatography-Tandem Mass Spectrometry (LC-MS/MS)
Gut and host microbiota-derived metabolites (III) | Before and after (12 weeks) of the intervention
  Changes in circulating succinate levels [µM]; assesed by EnzyChrom™ Succinate Assay Kit
Entero-endocrine incretin hormones (I) | Before and after (12 weeks) of the intervention
  Changes in post-prandial response to a meal-tolerance test in serum levels of glucose [mg/dL]; assesed by ELISA kit
Entero-endocrine incretin hormones (II) | Before and after (12 weeks) of the intervention
  Changes in post-prandial response to a meal-tolerance test in serum levels of insulin levels [pmol/L] ]assesed by ELISA kit
Entero-endocrine incretin hormones (III) | Before and after (12 weeks) of the intervention
  Changes in post-prandial response to a meal-tolerance test in plasma levels of glucagon-like peptite 1 [GLP-1 ] (pmol/L); assesed by ELISA kit
Entero-endocrine incretin hormones (IV) | Before and after (12 weeks) of the intervention
  Changes in post-prandial response to a meal-tolerance test in plasma levels of gastric inhibitory polypeptide (GIP) [pg/mL]; assesed by ELISA kit
Microbial composition/metagenomic | Before and after (12 weeks) of the intervention
  Changes in alpha and beta diversity, relative abundance and functional metagenomics; assesed by Ilumina metagenomics
Cellular energy metabolism | Before and after (12 weeks) of the intervention
  Changes in Cluster of Differentiation 14 positive (CD14+) monocytes isolated from peripheral blood mononuclear cells (PBMCs) will be used for bioenergetics analysis via an extracellular flux analyzer

CONTACTS AND LOCATIONS:
Overall Officials: Juan José Vendrell Ortega, Professor, Principal Investigator — Instituto de Investigación Sanitaria Pere Virgili (IISPV)
Locations (1):
- Hospital Universitario de Tarragona Juan XXIII, Tarragona, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No